CLINICAL TRIAL: NCT05127590
Title: A Phase 1b/2, Multicenter, Single Arm Study of RBN-2397 in Combination With Pembrolizumab in Patients With Squamous Cell Carcinoma of the Lung (SCCL)
Brief Title: RBN-2397 in Combination With Pembrolizumab in Patients With SCCL
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ribon Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RBN-2397-21-002
Record Dates: First submitted 2021-11-04; First posted 2021-11-19 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Advanced Squamous Non-Small Cell Lung Carcinoma
Keywords: NSCLC; Squamous Cell Lung Cancer; Squamous - NSCLC
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: RBN-2397 in combination with pembrolizumab
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RBN-2397 in combination with pembrolizumab (Experimental): RBN-2397 orally in combination with the fixed approved dose of IV pembrolizumab
  Interventions: Drug: RBN-2397

INTERVENTIONS:
Drug: RBN-2397 — Continuous oral dosing with the RP2D of RBN-2397 (outpatient basis). Pembrolizumab IV infusion over 30 minutes in clinic on Day 1 of each cycle.
  Other Names: Pembrolizumab; Keytruda

SUMMARY:
RBN-2397 inhibits PARP7, an enzyme that is switched on by cancer stresses, such as the toxins in cigarette smoke. Cancer cells use PARP7 to hide from the immune system by stopping the cell from sending a signal (Type 1 interferon) that tells the immune system that something is wrong and to kill the cell. RBN-2397 has been shown in animal and human studies to inhibit tumor growth and also shuts down the "don't kill me" signal the tumor is sending to evade the immune system.

The purpose of this study is to determine if RBN-2397 in combination with pembrolizumab (a PD-1 inhibitor) has the ability to restore the response to treatment in patients with SCCL that have been previously treated with a PD-1/PD-1 ligand (PD-L1) inhibitor and have had a response followed by disease progression.

The Phase 1b portion of the study will assess the safety of RBN-2397 in combination with pembrolizumab (a PD-1 inhibitor) and define the dose of RBN-2397 to be used in combination with pembrolizumab for the Phase 2.

The Phase 2 portion of the study will assess the anti-tumor activity of RBN-2397 in combination with pembrolizumab.

DETAILED DESCRIPTION:
This is an open label, multicenter Phase 1b/2 single arm study that will evaluate the safety and antitumor activity of RBN-2397 in combination with pembrolizumab in patients with confirmed diagnosis of advanced squamous cell carcinoma of the lung who have received prior therapy. The study consists of a Phase 1b Safety Run in and Phase 2.

During the Phase 1b Safety Run-in, approximately 10 patients will be enrolled in a 3+3 fashion and treated with continuous oral dosing with RBN-2397 twice daily (BID) in combination with the fixed approved dose of intravenous (IV) pembrolizumab every 3 weeks [Q3W]) to establish RP2D of RBN-2397 in combination with pembrolizumab.

During Phase 2, approximately 40 patients will be treated with continuous oral dosing with the RP2D of RBN-2397 BID in combination with the fixed approved dose of IV pembrolizumab.

In both the Phase 1b Safety Run in and Phase 2, a treatment cycle is defined as 21 days. On Day 1 of each treatment cycle, RBN-2397 will be administered orally and followed by IV infusion of pembrolizumab at the fixed approved dose according to the approved local product label. During the remaining days of the 21-day treatment cycle, only RBN-2397 BID will be administered. Treatment cycles will continue until disease progression, unacceptable treatment-related toxicity, or withdrawal of consent

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of advanced/metastatic NSCLC of squamous cell histology as determined by local testing practices.
2. Patients should have received prior therapy including a platinum containing chemotherapy regimen and an ICI, including anti-PD-1/anti-PD-L1, anti-cytotoxic T-lymphocyte-associated antigen 4 (CTLA-4) inhibitors, either sequentially or as combination of chemo + checkpoint inhibitor.
3. The last regimen prior to enrolling in the study must be a checkpoint inhibitor-containing regimen where the best response for at least one tumor response assessment was stable disease (SD), partial response (PR), or complete response (CR).
4. Patients experienced PD as determined by the investigator during or following their most recent treatment regimen
5. Must agree to undergo tumor biopsy if medically safe and feasible. Archival biopsy samples may be submitted if fresh biopsy can't be obtained.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
7. CT or MRI imaging done within 28 days prior to study treatment and have at least one measurable target lesion
8. Normal organ and bone marrow function
9. Patient and his/her partner agree to use adequate contraception during and for 3 months after the last study drug dose

Exclusion Criteria:

1. Has non-squamous histology NSCLC. Patients whose tumors have a mixed histology are ineligible.
2. Patient should not have received more than two prior lines of therapy with ICI including anti-PD-1/anti-PD-L1, anti-CTLA-4 inhibitors and one prior line of a chemotherapy treatment.
3. Patient is unable to swallow oral medications, has impairment of gastrointestinal (GI) function or GI disease that may significantly alter drug absorption (e.g., active inflammatory bowel disease, uncontrolled nausea, vomiting, diarrhea, or malabsorption syndrome).
4. Prior radiation within 2 weeks of Cycle 1 Day 1 (C1D1), except for palliative radiotherapy to a limited field. Patients must have recovered from all radiation related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤ 2 weeks of radiotherapy) to non CNS disease.
5. A patient with CNS metastases is excluded if:

   * Has active CNS metastases (new lesions or progression from prior imaging study) requiring treatment within 28 days prior to study treatment and/or ongoing corticosteroid therapy.
   * Has symptomatic or untreated leptomeningeal disease.
6. Patients who discontinue prior treatment with an ICI due to irAEs.
7. Has a known history of prior malignancy within the last 5 years. Except: malignancies that were treated curatively and have not recurred within 2 years prior to study treatment; completely resected basal cell and squamous cell skin cancers; any malignancy considered to be indolent and that has never required therapy; and completely resected carcinoma in situ of any type.
8. Has received a live-virus vaccination within 30 days of planned treatment start. Vaccines that do not contain live virus are permitted.
9. Any of the following in the previous 6 months: myocardial infarction or current history of New York heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular anemias, or electrocardiographic evidence of acute ischemia.
10. Patient has a history of prolonged QT syndrome or Torsades de pointes, and/or has a familial history of prolonged QT syndrome.
11. Patient is taking a concomitant medication that is a strong inhibitor or inducer of cytochrome P450 [CYP]-mediated metabolism or that is metabolized by CYP 2B6, 3A4 or 2C19, 2C9, or other members of the IIC subfamily of the CYP genes and that, if underdosed, would constitute a significant risk to the patient. Individual cases may be discussed with the Medical Monitor.
12. Ingestion of herbal medicines and grapefruit, grapefruit juice, pomegranate juice, star fruit, or orange marmalade (made with Seville oranges) from the start of the screening period. (Note that there are well- reported cases of CYP3A drug-drug interactions with these foodstuffs.)
13. Has active autoimmune disease that has required systemic treatment in the past 12 months (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., ≤ 10 mg daily prednisolone or steroid equivalent, thyroxine, insulin, or corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Patients with vitiligo, resolved childhood asthma/atopy, type I diabetes mellitus, and residual hypothyroidism due to an autoimmune condition and only requiring hormone replacement, are not excluded.
14. Is on chronic systemic steroids (e.g., > 10 mg daily prednisolone or steroid equivalent for > 6 months). Subjects with asthma that require intermittent use of bronchodilators, inhaled steroids, or local steroid injections would not be excluded from the study.
15. Has an active systemic infection requiring therapy (e.g.: bacterial, fungal, viral).
16. Has known active Hepatitis B or C. Active Hepatitis B is defined as a known positive HBsAg result. Active Hepatitis C is defined by a known positive Hepatitis C Antibody result and known quantitative hepatitis C virus ribonucleic acid (RNA) results greater than the lower limits of detection of the assay.
17. Has known psychiatric or substance abuse disorder that would interfere with cooperation with the requirements of the trial.
18. Has interstitial lung disease or a history of pneumonitis that required oral or intravenous steroids to assist with management. Lymphangitic spread of the NSCLC is not exclusionary.
19. Is pregnant or breastfeeding or expecting to conceive or father children while on study medication and for the required duration of contraception after the last dose of study medication.
20. Has ongoing acute clinical AEs of National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Grade ≥2 resulting from prior cancer therapies (except alopecia, peripheral neuropathy and ototoxicity, which are excluded if ≥ Grade 3).
21. Has had, within the past 6 months, the occurrence of one or more of the following events: cerebrovascular accident, deep vein thrombosis, pulmonary embolism, hemorrhage (CTCAE Grade 3 or 4), chronic liver disease (meeting criteria for Child Pugh Class B or C), organ transplantation.
22. Has, within 2 weeks prior to Day 1, received systemic therapeutic doses of corticosteroids (e.g., > 10 mg daily prednisolone or steroid equivalent). Topical, inhaled, nasal and ophthalmic steroids are allowed for short term treatment of acute conditions (e.g.: asthma, poison ivy contact dermatitis); for other immunosuppressive agents, the exclusionary dose and duration will be determined in consultation with the Medical Monitor.
23. Has any other medical or personal condition that, in the opinion of the Investigator, may potentially compromise the safety or compliance of the patient, or may preclude the patient's successful completion of the clinical study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Determine recommended Phase 2 dose (RP2D) (Phase 1b) | through study completion (an average of 6 months)
  Incidence rate of Dose limiting Toxicities (DLTs) of RBN 2397 in combination with pembrolizumab
Overall Response Rate (Phase 2) | From start of treatment (C1D1) up to 78 weeks
  Proportion of patients with confirmed response of CR or PR (RECIST v1.1)

SECONDARY OUTCOMES:
Safety determined by Treatment-Emergent Adverse Events | From start of treatment through 90 days after the last dose of study drug
  Incidence and severity of adverse events/serious adverse events as assessed by NCI CTCAE, version 5.0
Cmax of RBN-2397 | Through Study Day 22
  Assessment of Maximum plasma concentration (Cmax)
Tmax of RBN-2397 | Through Study Day 22
  Time to maximum plasma concentration (Tmax)
AUC of RBN-2397 | Through Study Day 22
  Assessment of area under the curve (AUC) of RBN-2397
T1/2 of RBN-2397 | Through Study Day 22
  Assessment of terminal half-life (T1/2) of RBN-2397

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Johnson, MD, Principal Investigator — Tennessee Oncology
Locations (19):
- United States (4):
  - Helen F. Graham Cancer Center (Christiana Care), Newark, Delaware
  - Cancer Treatment Centers of America, Newnan, Georgia
  - Hematology and Oncology Clinic, Baton Rouge, Louisiana
  - Sarah Cannon Research Institute, Nashville, Tennessee
- Israel (3):
  - Rambam Care Campus, Haifa
  - Hadassah Medical Center, Jerusalem
  - Shaare Zedek Medical Center, Jerusalem
- Spain (8):
  - Hospital Clinico Universitario De Santiago De Compostela, A Coruña
  - NEXT Oncology Barcelona, Barcelona
  - Vall D'Hebron Insitute of Oncology, Barcelona
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Quiron Madrid, Pozuelo de Alarcón
  - Hospital Universitario Virgen Macarena, Seville
  - INCLIVA Biomedical Research Institute, Valencia
- United Kingdom (4):
  - Beatson West of Scotland Cancer Centre, Glasgow, Scotland
  - Imperial College London, London
  - Sarah Cannon Research Institute UK (University College London Hospitals), London
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cohen MS, Chang P. Insights into the biogenesis, function, and regulation of ADP-ribosylation. Nat Chem Biol. 2018 Feb 14;14(3):236-243. doi: 10.1038/nchembio.2568. PMID 29443986
- [Background] Gozgit JM, Vasbinder MM, Abo RP, Kunii K, Kuplast-Barr KG, Gui B, Lu AZ, Molina JR, Minissale E, Swinger KK, Wigle TJ, Blackwell DJ, Majer CR, Ren Y, Niepel M, Varsamis ZA, Nayak SP, Bamberg E, Mo JR, Church WD, Mady ASA, Song J, Utley L, Rao PE, Mitchison TJ, Kuntz KW, Richon VM, Keilhack H. PARP7 negatively regulates the type I interferon response in cancer cells and its inhibition triggers antitumor immunity. Cancer Cell. 2021 Sep 13;39(9):1214-1226.e10. doi: 10.1016/j.ccell.2021.06.018. Epub 2021 Jul 22. PMID 34375612